CLINICAL TRIAL: NCT02980952
Title: Amino Acid Balance During Physical Inactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 157758/03
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Assessing Muscle Amino Acid Balance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy-balanced diet (Placebo Comparator): Forearm immobilization whilst consuming an energy-balanced diet
  Interventions: Other: Forearm immobilization
- High-fat overfeeding (Experimental): Forearm immobilization whilst consuming a high-fat diet, 50% energy excess
  Interventions: Other: High-fat overfeeding; Other: Forearm immobilization

INTERVENTIONS:
Other: High-fat overfeeding
  Arms: High-fat overfeeding
Other: Forearm immobilization

SUMMARY:
The aim is to assess the impact of physical inactivity on muscle amino acid balance and forearm glucose uptake. In addition, we will evaluate how high-fat overfeeding will modulate muscle amino acid balance and forearm glucose uptake.

DETAILED DESCRIPTION:
The aim is to assess the impact of forearm cast immobilization on muscle amino acid balance and forearm glucose uptake. In addition, we will evaluate how high-fat overfeeding during immobilization will modulate muscle amino acid balance and forearm glucose uptake.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes).
* Any diagnosed cardiovascular disease or hypertension.
* Elevated blood pressure at the time of screening. (An average systolic blood pressure reading of ≥140 mmHg over two or more measurements and an average diastolic blood pressure of ≥90 mmHg over two or more measurements.)
* Chronic use of any prescribed or over the counter pharmaceuticals.
* Regular use of nutritional supplements (e.g. creatine, protein supplementation)
* Metallic implants (including heart pacemaker, cochlear implants, medication pumps, surgical clips, plates or screws).
* A personal or family history of thrombosis, epilepsy, seizures or schizophrenia.
* Any previous motor disorders.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Muscle amino acid balance | 3 hours
  Forearm muscle amino acid balance

SECONDARY OUTCOMES:
Glucose uptake | 3 hours
  Forearm glucose uptake

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Wall, PhD, Principal Investigator — University of Exeter

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wall BT, Cruz AM, Otten B, Dunlop MV, Fulford J, Porter C, Abdelrahman DR, Stephens FB, Dirks ML. The Impact of Disuse and High-Fat Overfeeding on Forearm Muscle Amino Acid Metabolism in Humans. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa184. doi: 10.1210/clinem/dgaa184. PMID 32303743
- [Derived] Dirks ML, Wall BT, Otten B, Cruz AM, Dunlop MV, Barker AR, Stephens FB. High-fat Overfeeding Does Not Exacerbate Rapid Changes in Forearm Glucose and Fatty Acid Balance During Immobilization. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz049. doi: 10.1210/clinem/dgz049. PMID 31609422